CLINICAL TRIAL: NCT07247019
Title: The Effectiveness of Mobile Application Prototype (NutriDent4Mom) in Improving Nutrient Intake, Diet Quality, and Periodontal Health Status of Pregnant Women: A Cluster Randomized Trial
Brief Title: Effectiveness NutriDent4Mom to Improve Nutrient Intake, Diet Quality, and Periodontal Health Status of Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORKHAFIZAH SADDKI (Other)
Responsible Party: Sponsor-Investigator, NORKHAFIZAH SADDKI, ASSOCIATE PROFESSOR DR., Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USM/JEPeM/22020106
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Periodontal Disease; Nutrient Intake; Diet Quality
Keywords: pregnant women; periodontal health; nutrient intake; diet quality; mobile application
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NutriDent4Mom application (Experimental): NutriDent4Mom mobile application provides comprehensive nutrition and oral health education with attractive application features that enable the engagement of behavioral changes in nutrient intake and oral health care
  Interventions: Behavioral: Mobile Application Prototype
- Ministry of Health healthcare program for antenatal mothers (Active Comparator): Routine antenatal healthcare provided by the MOH staff which include delivery of health education according to the topics specified in the Antenatal Mother Record Book or "Buku Rekod Kesihatan Ibu"
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Mobile Application Prototype — Participants were provided with the NutriDent4Mom application installed in their own mobile device. They were instructed to use the apps throughout the study period. The instructions include entering the daily food intake and reading the educational content. The participants must finish reading the content, which covers at least two topics per day, within one week. The mobile application usage was monitored by a usage counter, and participants also received reminders to record their diet intake into the application.
  Arms: NutriDent4Mom application
Behavioral: Health education — Participants received health education delivered via health talk. Oral health care is one of the topics among other health topics including diet, breastfeeding, family planning, and preparation for delivery. These health education topics were delivered by the MOH medical staff nurses except for oral health care which was delivered by dental officers.
  Arms: Ministry of Health healthcare program for antenatal mothers

SUMMARY:
The goal of this two-arm, parallel-group cluster randomized controlled trial was to assess the effectiveness of a healthcare mobile application prototype (NutriDent4Mom) in improving nutrient intake, diet quality and periodontal health status of pregnant women.

The main questions it aims to answer are:

1. Does the NutriDent4Mom apps increase the mean nutrient intake (Nutrient value) and diet quality score (HEI) of pregnant women?
2. Does the NutriDent4Mom apps improve the periodontal health (GI score, CPI score) of pregnant women?

Researchers will compare the NutriDent4Mom apps to the conventional Ministry of Health (MOH) program to see if the NutriDent4Mom apps is effective to improve nutrient intake, diet quality and periodontal health status of pregnant women.

DETAILED DESCRIPTION:
Participants will receive the NutriDent4Mom application. Measurement of outcomes included the 3-day 24-hour diet recall for nutrient intake, Food Frequency Questionnaire (FFQ) for diet quality, and the Gingival Index (GI) and Community Periodontal Index (CPI) for periodontal health. Data were collected 3 times, at baseline before the respective intervention, after one month (evaluation 1), and after another one month (evaluation 2).

ELIGIBILITY:
Inclusion Criteria:

* Aged from 19 to 50 years old
* Pregnant between 13 to 20 weeks
* Singleton pregnancy
* Own any type of android operating system handheld device
* Malaysian citizen
* Able to read and write in Malay language

Exclusion Criteria:

* Diagnosed with diabetes mellitus or gestational diabetes mellitus
* Diagnosed with hypertensive disorder
* Diagnosed with severe hyperemesis gravidarum during current pregnancy
* Wearing dental appliances (removable and/or fixed appliance)

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study enrolled pregnant women. Therefore, only females are eligible to participate
Enrollment: 264 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Nutrient Value | From baseline to the end of intervention period at 8 weeks
  Nutrient intake was assessed using 24-hour diet recall. The 24-hour recall was done for 3 days (1 weekend and 2 weekdays) to establish intake of nutrients. Data were analysed using Nutritionist Pro™ software to establish the nutrient intake value. The nutrient values were compared with the Recommended Nutrient Intake (RNI) for pregnancy and categorised as follows: 1) Inadequate for values below the estimated average requirement, 2) Adequate for values between the estimated average requirement and tolerable upper intake level, and 3) Excessive for values exceed the tolerable upper intake level.
Healthy Eating Index | From baseline to the end of intervention period at 8 weeks
  Diet quality was assessed using a self-administered semi-quantitative food frequency questionnaire (FFQ). The FFQ comprises of 82 food items organized into 10 main food groups as follows: 1) Cereal and cereal products, 2) Meat and eggs, 3) Milk and milk products, 4) Nuts, 5) Vegetables, 6) Fruits and fruit juices, 7) Beverages, 8) Fats, 9) Sweet and baked goods, and 10) Condiments. The frequency of food intake has a 7-point scale rating as follows: 1=never or rarely, 2=once a month, 3=2 to 3 times a month, 4=once a week, 5=2 to 3 times a week, 6=once daily, and 7=2 to 3 times daily. The conversion factor was used to estimate food intake based on frequency of intake. The score of each food group was calculated using a validated formula. Diet quality was categorized as 1) Poor diet for score less than 51%, 2) diet requiring improvement for score 51 to 80%, and 3) Good diet for score more than 80%.
Mean Gingival Index score | From baseline to the end of intervention period at 8 weeks
  The Gingival Index (GI) was used to assess the severity of gingival inflammation. Four gingival areas of 6 index teeth (16, 12, 24, 36, 32 and 44) were examined using a CPI probe and given scores as follows: 0 = normal healthy gingiva; 1 = mild inflammation with slight colour change and oedema but no bleeding on probing; 2 = moderate inflammation with red, oedematous and glazing gingival tissues that bleed on probing; and 3 = severely inflamed gingival tissues with marked redness and oedema, ulceration, and tendency to bleed spontaneously. The scores from each index tooth were added and divided by 4 to give the GI for the tooth. The GI of each patient was determined by adding the scores for all index teeth and dividing it by the number of teeth examined.
Mean Community Periodontal Index score | From baseline to the end of intervention period at 8 weeks
  Periodontal health status was measured using the Community Periodontal Index (CPI). The mouth was divided into 6 sextants (18-14, 13-23, 24-28, 38-34, 33-43, 44-48) and 10 index teeth (17, 16, 11, 26, 27, 36, 37, 31, 47, and 46) were examined using a CPI probe and given scores as follows: 0 = healthy periodontium, 1 = bleeding after probing, 2 = calculus detected during probing but the black band on the probe was visible, 3 = shallow pocket 4-5 mm (gingival margin within the black band on the probe), and 4 = deep pocket ≥ 6 mm (black band on the probe not visible). The highest CPI score of each patient was recorded, and the mean number of sextants having CPI code of 0, 1, 2, 3, and 4 was calculated to indicate the severity of periodontal disease.

CONTACTS AND LOCATIONS:
Overall Officials: NORKHAFIZAH SADDKI, MCommMed (Oral Health) (USM), Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Ministry of Health Maternal and Child Health Clinics, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No
Ethical considerations